CLINICAL TRIAL: NCT00719108
Title: Randomized,Single Center,Double Blind,Two-period,Crossover Glucose Clamp Trial to Test Bioequivalence Between Two Recombinant Human Soluble Insulins - Wockhardt's Insulin Human Regular for Injection and Actrapid, in Healthy Subjects
Brief Title: Comparative Glucose Clamp Study of Wockhardt's Insulin Human Regular for Injection and Actrapid, in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: WosulinR/PK-PD/HV/EMEA/2008/v2
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Diabetes
Keywords: Diabetes, Healthy Volunteers
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wosulin R (Experimental): Wosulin R, Regular insulin for injection (Recombinant Human Insulin) (100 IU/mL)in vials 10.0 ml
  Interventions: Biological: Wosulin R
- Actrapid (Active Comparator): Actrapid, Regular insulin for injection (Recombinant Human Insulin) (100 IU/mL)in vials 10.0 ml
  Interventions: Biological: Actrapid

INTERVENTIONS:
Biological: Wosulin R — Total dose per subject will be 0.3 IU/Kg given IV over 5 hrs.
  Arms: Wosulin R
Biological: Actrapid — Total dose per subject will be 0.3 IU/Kg given IV over 5 hrs.
  Arms: Actrapid

SUMMARY:
The aim of this trial is to demonstrate bioequivalence of Wosulin R to Actrapid with regard to its total and to its maximum serum insulin concentrations.

DETAILED DESCRIPTION:
The purpose of this study is the comparative evaluation of the Pharmacodynamics and Pharmacokinetics of two recombinant regular human insulin injections administered intravenously in healthy volunteers under the conditions of euglycemic clamp.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subject
2. Age between 18 and 45 years (both inclusive)
3. Considered generally healthy upon completion of medical history, physical examination and biochemical investigations as judged by the Investigator.
4. Body Mass Index (BMI) between 18.0 and 35.0 kg/m2 (both inclusive)
5. Non-smoker, defined as no nicotine consumption for at least one year.
6. Signed and dated informed consent obtained before any trial-related activities.

Exclusion Criteria:

1. Previous participation in this trial or other clinical trials within the last 3 months.
2. Pregnant, breast-feeding or intention of becoming pregnant or not using adequate contraceptive measures.
3. Clinically significant abnormal hematology or biochemistry screening tests, as judged by the Investigator.
4. Any serious systemic infectious disease during the four weeks prior to the first dose of test drug, as judged by the Investigator.
5. History of any illness that, in the opinion of the Investigator, might confound the results of the trial or pose risk in administering the trial drug to the subject. In particular, subjects with significant cardiovascular disease, anemia (below the lower limit of normal) or hemoglobinopathy will not be allowed to enter the trial.
6. History of alcohol or drug abuse within the past 5 years and/or any positive test for drugs of abuse at screening.
7. Positive test for hepatitis B or C or HIV positive at screening or in the past.
8. Use of prescription drugs within 3 weeks preceding the first dosing of insulin, except for oral contraceptives/hormonal implants.
9. Use of any insulin product in the past.
10. Use of non-prescription drugs, except routine vitamins, within 2 weeks prior to the first dose of the test drug. Occasional use of acetaminophen will be permitted.
11. Blood donation of more than 500 mL (or considerable blood loss) within the last 12 weeks.
12. History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
13. Known or suspected allergy to trial products or related products.
14. Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The area under the GIR-time curve at steady state from 240 to 300 minutes (AUCGIR-SS) | Visit 2 and 3

SECONDARY OUTCOMES:
PD Endpoints: Area under the GIR-time curve from 0 to 7 hours, GlR at steady state. PK Endpoints: AUCINS-SS, AUCINS0-7h, CLtot, VSS, t1/2 ,Terminal rate constant Safety Endpoints: AE, Lab assessments, Vital signs, Phy Exam, ECG & Hypoglycemia. | Visit 2 , 3 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Hompesch, MD, Study Director — Profil Institute of Clinical Research
Locations (1):
- Profil Institute for Clinical Research Inc., Chula Vista, California, United States